CLINICAL TRIAL: NCT04707482
Title: Cohort Study of Mechanism and Process Regulation for Colorectal Tumors
Brief Title: Mechanism and Process Regulation for Colorectal Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government); RenJi Hospital (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: mechanism for CRC
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer; Adenoma
Keywords: Colorectal cancer; Adenoma; Mechanism; Process regulation
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue sample, blood sample, stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study focused on the key nodes, molecular events and regulatory mechanisms of intestinal microecological disorders that affect the malignant transformation of intestinal epithelial cells into tumors during the occurrence and development of colorectal cancer.

DETAILED DESCRIPTION:
Phase Ⅰ is a cross-sectional study to record selected information and biospecimen of more than 250 sporadic colorectal adenoma cases (200 cases with convetional adenomas, 25 cases with hyperplasticpolyps and 25 cases with TSA/SSAs), 50 cases of sporadic colorectal cancer (early cancer), 50 cases with familial inherited colorectal cancer (FAP and LS) or healthy controls.

Phase Ⅱ is a nested case-control study. A total of 250 patients with sporadic colorectal cancer (early stage cancer) or sporadic colorectal adenoma will be included in Phase Ⅱ and regular follow-up to observe the recurrence and progress after resection of the lesions of colorectal adenomas.

The end point of the study is the recurrence of bowel adenoma or carcinoma and follow-up time is five years. After the observation, each case with the study outcome was matched with corresponding controls in a 1:1 ratio for further analysis according to the conditions such as age and gender.(Due to the particularity of single-cell sequencing, all specimens that meet the test requirements were sent for examination, and a nest-type case-control design was not adopted.)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria（Healthy control group）： 1) Aged more than 18 years; 2) Planned to undergo colonoscopy , without past medical history of neoplasm or ulcer or bleeding under colonoscopy regardless of the history of colonoscopy; 3) Willing to participate in this trial and signed the informed consent.

  * Inclusion Criteria（Sporadic colorectal adenoma group）：

    1. More than 18 years aged;
    2. Diagnosed as colorectal adenoma, epithelial adenomatoid hyperplasia, serrated lesions, or with mild to moderate dysplasia (low-grade intraepithelial neoplasia) by colonoscopy and pathology;
    3. Signed the informed consent, willing to participate in this trial.
  * Inclusion Criteria（Sporadic early colorectal cancer group）：

    1. Aged more than 18 years;
    2. Underwent endoscopic EMR/ESD or Surgical resection because of colorectal neoplasms and the lesion was confined to the mucosa or submucosa of the large intestine and was pathologically indicated to be adenocarcinoma;
    3. Willing to participate in this trial and signed the informed consent.
  * Inclusion Criteria（Familial colorectal neoplasm group）：

    1. Aged more than 18 years;
    2. Underwent ESD/EMR resection or surgical resection and the pathology result considered as early colorectal cancer and adenoma, and the family history, pathology and genetic tests met the diagnostic criteria of FAP and HNPCC/LS;
    3. Signed the informed consent, willing to participate in this trial. ·-Inclusion Criteria (Cohort study)

    <!-- -->

    1. Aged 18-80 years;
    2. Diagnosed as polypoid neoplasm or lateral developmental neoplasm (LST) by endoscopy without a family history of CRC and the pathologic manifestations were conventional adenoma or serrated lesions; the patients without a family history of CRC underwent ESD or EMR resection and the pathology result considered as early colorectal cancer; diagnosed as sporadic colorectal early carcinoma and adenoma with a family history of colorectal cancer (FAP, Lynch syndrome);
    3. Signed the informed consent, willing to participate in this study and agreed with colonoscopy with pathology examination once a year and followed up for 5 years.

Exclusion Criteria:

* -Exclusion Criteria（Healthy control group）：

  1. With a medical history of digestive tract rerouting and partial resection;
  2. Patients with high risk of hereditary colorectal adenocarcinoma, i.e. family members of the following diseases: family history of gastrointestinal neoplasms, familial adenomatous polyposis (FAP), hereditary non-polyposis colorectal adenocarcinoma (HNPCC/LS), and P-J syndrome;
  3. With A history of chronic metabolic and inflammatory diseases such as hypertension, diabetes, chronic viral hepatitis, and inflammatory bowel disease and the chronic disease were difficult to control;
  4. With other malignancies known to have advanced or require treatment in the past 5 years, except basal cell and squamous cell carcinoma of the skin that have been radically cured;
  5. With a history of active gastrointestinal bleeding within the last 6 months;
  6. With a history of using broad-spectrum antibiotics and probiotics by oral or intravenous within the past 1 month;
  7. Received routine immunosuppressive drugs for the past 6 months;
  8. Unable or unwilling to cooperate with follow-up and related examinations;
  9. Patients who can not eat normally or need to rely on medicine or enema and other defecation;
  10. With mental illness or any other serious cardiovascular disease;
  11. With pregnant or lactating or planning to become pregnant within one year;
  12. Currently participating in, or receiving, an interventional clinical study that affects patients' treatment decisions.
* Exclusion Criteria（Sporadic colorectal adenoma group）：

  1. With a medical history of digestive tract rerouting and partial resection;
  2. Patients with high risk of hereditary colorectal adenocarcinoma, i.e. family members of the following diseases: family history of gastrointestinal neoplasms, familial adenomatous polyposis (FAP), hereditary non-polyposis colorectal adenocarcinoma (HNPCC/LS), and P-J syndrome;
  3. With A history of chronic metabolic and inflammatory diseases such as hypertension, diabetes, chronic viral hepatitis, and inflammatory bowel disease and the chronic disease were difficult to control;
  4. With other malignancies known to have advanced or require treatment in the past 5 years, except basal cell and squamous cell carcinoma of the skin that have been radically cured;
  5. With a history of active gastrointestinal bleeding within the last 6 months;
  6. With a history of using broad-spectrum antibiotics and probiotics by oral or intravenous within the past 1 month;
  7. Received routine immunosuppressive drugs for the past 6 months;
  8. Unable or unwilling to cooperate with follow-up and related examinations;
  9. Patients who can not eat normally or need to rely on medicine or enema and other defecation;
  10. With mental illness or any other serious cardiovascular disease;
  11. With pregnant or lactating or planning to become pregnant within one year;
  12. Currently participating in, or receiving, an interventional clinical study that affects patients' treatment decisions.
* Exclusion Criteria（Sporadic early colorectal cancer group）：

  1. With a medical history of digestive tract rerouting and partial resection;
  2. Patients with high risk of hereditary colorectal adenocarcinoma, i.e. family members of the following diseases: family history of gastrointestinal neoplasms, familial adenomatous polyposis (FAP), hereditary non-polyposis colorectal adenocarcinoma (HNPCC/LS), and P-J syndrome;
  3. With A history of chronic metabolic and inflammatory diseases such as hypertension, diabetes, chronic viral hepatitis, and inflammatory bowel disease and the chronic disease were difficult to control;
  4. With other malignancies known to have advanced or require treatment in the past 5 years, except basal cell and squamous cell carcinoma of the skin that have been radically cured;
  5. With a history of active gastrointestinal bleeding within the last 6 months;
  6. With a history of using broad-spectrum antibiotics and probiotics by oral or intravenous within the past 1 month;
  7. Received routine immunosuppressive drugs for the past 6 months;
  8. Unable or unwilling to cooperate with follow-up and related examinations;
  9. Patients who can not eat normally or need to rely on medicine or enema and other defecation;
  10. With mental illness or any other serious cardiovascular disease;
  11. With pregnant or lactating or planning to become pregnant within one year;
  12. Currently participating in, or receiving, an interventional clinical study that affects patients' treatment decisions.
* Exclusion Criteria（Familial colorectal neoplasm group）：

  1. With a medical history of digestive tract rerouting and partial resection;
  2. With A history of chronic metabolic and inflammatory diseases such as hypertension, diabetes, chronic viral hepatitis, and inflammatory bowel disease and the chronic disease were difficult to control;
  3. With a history of active gastrointestinal bleeding within the last 6 months;
  4. With a history of using broad-spectrum antibiotics and probiotics by oral or intravenous within the past 1 month;
  5. Received routine immunosuppressive drugs for the past 6 months;
  6. Unable or unwilling to cooperate with follow-up and related examinations;
  7. Patients who can not eat normally or need to rely on medicine or enema and other defecation;
  8. With mental illness or any other serious cardiovascular disease;
  9. With pregnant or lactating or planning to become pregnant within one year;
  10. Currently participating in, or receiving, an interventional clinical study that affects patients' treatment decisions.

      * Exclusion Criteria（Cohort study）

Except baseline exclusion criteria, and the following conditions should be excluded:

1. Diagnosed as advanced colorectal cancer (with or without surgery, radiation, chemotherapy, targeted therapy, immunotherapy);
2. Refuse to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal adenoma; early colorectal cancer; familial genetic colorectal cancer who underwent colonoscopy and met diagnostic criteria; healthy controls group
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Difference of bacteria species | May 1, 2022
  Difference of bacteria species between the recurrent and non recurrent colorectal adenomas.
Difference of metabolites of intestinal pathogenic bacteria | May 1, 2022
  Difference of metabolites of intestinal pathogenic bacteria between the recurrent and non recurrent colorectal adenomas.
Difference of immune markers | May 31, 2023
  Difference of immune markers between the recurrent and non recurrent colorectal adenomas.
Difference of protein expression | May 31, 2023
  Difference of protein expression between the recurrent and non recurrent colorectal adenomas.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Jing, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Ruijin Hospttal, Shanghai, Sahgnhai, China